CLINICAL TRIAL: NCT00624988
Title: The Effect of Vibration Therapy on the Bone Density of the Tiba in Patients With Spinal Cord Injury
Acronym: SCI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: David Lenihan BA., D.C., Ph.D., M.C.C., CBiol MiBiol, FRSM, Logan University, College of Chiropractic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD0723070100
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injury; vibration therapy; bone density
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vibration Therapy (Experimental): Treatment will consist of 10 sessions of 60 seconds each with one minute intervals in between at 50 Hz frequency three times per week for three months.
  Interventions: Procedure: Vibration Therapy

INTERVENTIONS:
Procedure: Vibration Therapy — Treatment will consist of 10 sessions of 60 seconds each with one minute intervals in between at 50 Hz frequency three times per week for three months.

SUMMARY:
The purpose of this investigation is to determine the effect of lower limb vibration therapy on bone density in the tibia in patients with spinal cord injury. The second purpose is to assess the neuromuscular junction variability at the motor units of the tibialis anterior muscle after a sequence of lower limb vibration therapy

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* A spinal cord injury patient with injury above T12
* Injury below T4 to avoid respiratory complication.
* An ASIA classification of A or B

Exclusion Criteria:

* Non complicating organic factors such as heart disease, high blood pressure, stroke
* Exercise where electrical therapy is used while the trial is being conducted
* A bone density measure 3 times below normal mineralization levels as measured on the first bone density scan prior to entry in to the study
* Surgical implants below the level of T12
* Local infection, acute inflammation, injury, tumors or other malignancy, recent wounds, diabetes
* Any unstable joints of the lower extremity, recent hip and knee joints or fitted hip or knee pins, bolts and/or plates
* Acute thrombosis
* Severe migraine, epilepsy
* Serious cardiovascular disease, wearing a pacemaker
* Any Spinal manipulation within one year of the study
* Any implanted device or prosthesis or intrauterine IUD type of device pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Bone density scan | within 7 days pre/post intervention

SECONDARY OUTCOMES:
Single fiber EMG at neuromuscular junction | 7 days pre/post intervention

CONTACTS AND LOCATIONS:
Overall Officials: David V Lenihan, DC, PhD, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States